CLINICAL TRIAL: NCT05967416
Title: Phase 1 Study of Autologous SIRPα-low Macrophages (SIRPant-M) Administered by IT- Injection Alone or in Combination With Focal External-Beam Radiotherapy in Participants With Relapsed or Refractory Non-Hodgkin's Lymphoma
Brief Title: Study of SIRPant-M in Participants With Relapsed or Refractory Non-Hodgkin's Lymphoma
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: SIRPant Immunotherapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SIRP01-1001
Record Dates: First submitted 2023-07-21; First posted 2023-08-01 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Refractory Non-Hodgkin Lymphoma; Relapsed Non-Hodgkin Lymphoma
Keywords: Non-Hodgkin Lymphoma; Relapsed/Refractory Non-Hodgkin Lymphoma; Autologous cell therapy
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Intervention Model Description: Enrollment will begin with Cohort 1, Group 1 (SIRPant-M monotherapy, low dose). Upon approval from the SRC after Cohort 1, Group 1 review, enrollment in Cohort 1, Group 2 (SIRPant-M coupled with XRT, low dose) and Cohort 2, Group 3 (SIRPant-M monotherapy, intermediate dose) will open. Upon approval from the SRC after Cohort 1, Group 2 and Cohort 2, Group 3 review, enrollment in Cohort 2, Group 4 (SIRPant-M + XRT, intermediate cell dose) will open. Upon further approval from the SRC, Cohort 3, Groups 5 and 6 (high cell dose + XRT, alternate day- versus weekly IT-dosing) will enroll.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- SIRPant-M (90×10^6 cells) (Experimental): SIRPant-M Monotherapy (Single Agent)
  Interventions: Biological: SIRPant-M
- SIRPant-M (90×10^6 cells) with focal XRT (Experimental): SIRPant-M coupled with 2.5 Gy of focal XRT administered within 24 hours after the first ITI and within 3 hours before to 24 hours after the second and third ITI
  Interventions: Biological: SIRPant-M; Radiation: External-beam radiotherapy (XRT)
- SIRPant-M (300×10^6 cells) (Experimental): SIRPant-M Monotherapy (Single Agent)
  Interventions: Biological: SIRPant-M
- SIRPant-M (300×10^6 cells) with focal XRT (Experimental): SIRPant-M coupled with 2.5 Gy of focal XRT administered within 24 hours after the first ITI and within 3 hours before to 24 hours after the second and third ITI
  Interventions: Biological: SIRPant-M; Radiation: External-beam radiotherapy (XRT)
- SIRPant-M (600×10^6 cells) with focal XRT, alternate Day 1, 3, 5 IT-dosing (Experimental): SIRPant-M coupled with 2.5 Gy of focal XRT administered within 24 hours after the first ITI and within 3 hours before to 24 hours after the second and third ITI
  Interventions: Biological: SIRPant-M; Radiation: External-beam radiotherapy (XRT)
- SIRPant-M (600×10^6 cells) coupled with focal XRT, weekly (W1, 2, 3) IT-dosing (Experimental): SIRPant-M coupled with 2.5 Gy of focal XRT administered within 24 hours after the first ITI and within 3 hours before to 24 hours after the second and third ITI
  Interventions: Biological: SIRPant-M; Radiation: External-beam radiotherapy (XRT)

INTERVENTIONS:
Biological: SIRPant-M — Autologous activated macrophage cell therapy manufactured from peripheral blood mononuclear cells given by intratumoral injection
Radiation: External-beam radiotherapy (XRT) — Radiotherapy given by external beam to the IT-injected lesion only
  Arms: SIRPant-M (300×10^6 cells) with focal XRT; SIRPant-M (600×10^6 cells) coupled with focal XRT, weekly (W1, 2, 3) IT-dosing; SIRPant-M (600×10^6 cells) with focal XRT, alternate Day 1, 3, 5 IT-dosing; SIRPant-M (90×10^6 cells) with focal XRT

SUMMARY:
The goal of this study is to test SIRPant-M (RB-1355) , an autologous cell therapy, alone or in combination with focal external-beam radiotherapy in participants with relapsed or refractory non-Hodgkin's lymphoma (NHL). Two dose levels of SIRPant-M are being tested. The main question this study aims to answer is if SIRPant-M alone or in combination with radiotherapy is safe and well-tolerated.

DETAILED DESCRIPTION:
This is an open-label phase 1 study of SIRPant-M studied in serial cohorts either alone (monotherapy), or combined with low-dose focal external-beam radiotherapy (XRT) in patients with relapsed- or refractory Non-Hodgkin's lymphoma (NHL). Both B-cell and certain T-cell NHL (select PTCL; CTCL) are eligible. The primary objective of the study is to assess the safety and tolerability of autologous SIRPant-M, delivered by 3 intra-tumoral injection, given either alone or combined with 2.5 Gy focal XRT.

A course (cycle) of SIRPant-M (RB-1355) is prepared from a single mononuclear apheresis, and comprises 3 equal ITI doses, administered at 2-day intervals. A low dose (90x10^6 cells split over 3 injections), an intermediate dose (300x10^6 cells split over 3 injections) and a high dose (600x10^6 cells split over 3 injections) of SIRPant-M are evaluated. In cohorts receiving supplemental radiation, each cell injection will be followed by 2.5 Gy radiation directed at the injected tumor site (7.5 Gy total). At the highest dose level only, alternate day IT-dosing (Day 1, 3, 5) will be compared with Weekly IT-dosing (W1, 2, 3).

Patients with PR or sustained clinical benefit (at least SD) after 1 cycle may receive a 2nd cycle of treatment, using cells prepared and frozen following the initial apheresis.

Dose escalations will be staggered using the 3+3 Phase 1 design, and safety will be monitored by the Safety Review Committee (SRC). The SRC may direct additional- or intermediate dose levels to be evaluated, as guided by emerging data.

ELIGIBILITY:
Inclusion Criteria:

1. Adult, defined as age ≥ 18 (at screening), who are willing and able to provide informed consent
2. Must have relapsed/refractory lymphoma, received at least 2 lines of systemic therapy, be ineligible or inappropriate for other treatment regimens known to have curative potential, and must have recovered from the acute toxic effects of all prior oncologic therapy of curative intent (except alopecia)
3. Histologically or cytologically confirmed diagnosis of NHL, any one of the below:

   1. Eligible for SIRPant-M monotherapy or SIRPant-M plus focal XRT combination therapy: Diffuse large B-cell lymphoma and cutaneous T-cell lymphoma (CTCL), including mycosis fungoides (MF), Sezary Syndrome, anaplastic large cell lymphoma (ALCL), lymphomatoid papulosis; adult T-cell leukemia/lymphoma (ATLL); peripheral T cell lymphoma; and angioimmunoblastic T cell lymphoma
   2. Eligible for SIRPant-M monotherapy only: Cutaneous B-cell lymphoma, including primary cutaneous follicle center lymphoma and primary cutaneous marginal zone B-cell, leg type; follicular center lymphoma; chronic lymphocytic leukemia (CLL) /small lymphocytic lymphoma (SLL); mantle cell lymphoma (MCL); nodal marginal zone B-cell lymphoma
4. Must have at least one accessible lymph node or cutaneous or subcutaneous lesion of 1.5 to 5 cm in one dimension as measured by computed tomography (CT) or positron emission tomography/computed tomography (PET/CT) or ultrasound for ITI by an interventional radiologist or other appropriately qualified and trained personnel, which presents a low risk for complications as determined by the Interventional Radiologist and the Principal Investigator. The target lesion must not have been previously irradiated. Note that lesions in the vicinity of large vessels, and tumor-encased large vessels are not considered low-risk. Additional caution should be taken in patients with neck lesions and lesions connected to ulcerated skin or mucosal surface. The target lesion must not be >5 cm in any dimension.
5. Must have a life expectancy > 3 months; must also be confirmed within 7 days prior to Day 1 of SIRPant-M ITI treatment
6. Must have an Eastern Cooperative Oncology Group (ECOG) Performance Status ≤ 2; must also be confirmed within 7 days prior to Day 1 of SIRPant-M ITI treatment
7. Must have hematologic values as follows: hemoglobin (Hgb) > 8 g/dL, ANC > 500 /mm3, monocyte counts ≥ 200/μL, and platelets > 50,000/µL; must also be confirmed within 7 days prior to Day 1 of SIRPant-M ITI treatment
8. Must have adequate renal and hepatic function as follows:

   1. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) <3× the upper limit of normal (ULN) (unless attributed to leukemic involvement or required concomitant medication)
   2. Calculated creatinine clearance ≥60 milliliter per minute (mL/min) calculated with Cockcroft-Gault formula
   3. Bilirubin ≤1.5×ULN, unless secondary to Gilbert's Syndrome.

   Must also be confirmed within 7 days prior to Day 1 of SIRPant-M ITI treatment.
9. Cardiac function: Must be American Heart Association (AHA) class 1 without significant limitation of physical activity; must also be confirmed within 7 days prior to Day 1 of SIRPant-M ITI treatment.
10. Must not be pregnant or planning to become pregnant. A negative urine or serum pregnancy test result is required for persons of reproductive potential within 72 hours prior to start of study treatment administration.
11. All persons of reproductive potential must agree to use an effective contraceptive method during study participation and for a minimum of 90 days after study treatment.

    1. Biologically female: is premenarcheal, surgically sterile (post hysterectomy, bilateral salpingectomy, or bilateral oophorectomy), postmenopausal (>12 months of amenorrhea without alternative medical causes), or, if of reproductive potential, is using a highly effective method of contraception (combined estrogen/progestogen or progestogen-only hormonal contraceptives associated with inhibition of ovulation, intrauterine device [IUD], intrauterine hormone-releasing system [IUS], bilateral tubal occlusion/ligation, vasectomized partner[s], double barrier method [male condom with either cap, diaphragm, or sponge with spermicide], or true abstinence of heterosexual intercourse when this is in line with the preferred and usual lifestyle of the person [periodic abstinence, eg, calendar, ovulation, symptom-thermal, post-ovulation methods, and withdrawal are not acceptable methods of contraception]), and agrees to continued use of this method until 90 days after end of study treatment
    2. Biologically male: is vasectomized and has received medical assessment of surgical success, has undergone bilateral orchidectomy, or agrees to use an approved method of contraception (true abstinence of heterosexual intercourse when this is in line with the preferred and usual lifestyle of the person, double barrier method [male condom with either cap, diaphragm, or sponge with spermicide], partner's use of a highly effective method of contraception sterile, partner is postmenopausal, or partner is surgically sterile) and agrees to use this method until 90 days after study treatment
12. In the opinion of the Investigator, must be willing and able to comply with the protocol for the duration of the study including undergoing treatment, the required tumor tissue biopsy procedures, scheduled visits and examinations, and including follow up

Exclusion Criteria:

1. Must not have received prior ITI therapy
2. Must not have received ASCT or treatment with cellular therapy including CAR-T within the prior 1 month; must not have received allogeneic stem cell transplantation within prior 6 months and must have no active graft-versus-host disease (GVHD) or be under active immunosuppression for GVHD.
3. Must not have received prior systemic anti-cancer therapy within the past 14 days before start of study cell therapy
4. Must not have received IL-2 therapy within the last 6 months
5. Must not have acquired immune defects such as human immunodeficiency virus (HIV)
6. Must not have uncontrolled hypertension (systolic >180 mmHg, diastolic >100 mmHg)
7. Must not have diagnosis of unclassifiable B cell lymphoma
8. Must not have bleeding diathesis or abnormal values for prothrombin time (PT) or activated partial thromboplastin time (aPTT), international normalized ratio (INR) > 1.5× ULN
9. Must not be receiving anti-platelet drugs that may present a risk for intratumor injections
10. Must not have pulmonary disease which, in the opinion of the Investigator, might impair the patient's respiratory tolerance to moderate pulmonary fluid overload (eg, interstitial lung disease, severe chronic obstructive pulmonary disease)
11. Must not have known alcohol or drug abuse
12. Must not have received an investigational agent within the past 30 days before start of study cell therapy
13. Must not require a chronic therapy with prednisone at a dose of or exceeding 10 mg/day or equivalent or any other form of immunosuppressive therapy
14. Must not have active central nervous system tumors or metastases
15. Must not be ineligible to receive 2.5 Gy ×3 focal external-beam radiation therapy as determined by the Radiation Oncologist and Principal Investigator (Cohort 1/Group 2, Cohort 2/Group 4, and Cohort -1/Group 4 only)
16. Must not have uncontrolled active viral hepatitis-B, -C, and/or -D infection
17. Must not have received a live vaccine within 4 weeks of the baseline/screening visit
18. Must not have active, uncontrolled autoimmune disease and/or history of autoimmune diseases at high risk for relapse
19. Must not have another malignancy or uncontrolled intercurrent illness, condition, serious medical or psychiatric illness, or circumstance that, in the opinion of the Investigator, could interfere with adherence to the study's procedures or requirements, or otherwise compromise the study's objectives
20. No active systemic infection; must also be confirmed on Day 1 prior to initiation of ITI

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-01-17 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of treatment emergent adverse events (TEAEs) and adverse events (AEs) | Day -42 through Day 364
  Includes evaluation of frequency and severity of AEs, serious adverse events (SAEs), TEAEs, and adverse events of special interest (AESIs), including injection site reactions and abnormalities in clinical laboratory assessments, vital signs, or physical examination findings. Graded according to Common Terminology Criteria for Adverse Events (CTCAE) Version 5.0.

SECONDARY OUTCOMES:
Recommended phase 2 dose of autologous SIRPant-M +/- 2.5 Gy ×3 focal XRT | Day 1 through Day 364
  Based on review of safety, pharmacodynamic, and efficacy data.
Objective response rate (ORR) | Day 1 through Day 364
  Based on number of participants with complete response (CR) and partial response (PR). Determined by positron emission tomography/computed tomography (PET/CT) and evaluated per the Lugano classification.

CONTACTS AND LOCATIONS:
Overall Officials: Jelle Kijlstra, MD, MBA, Study Director — BobcatBio, p/k/a SIRPant Immunotherapeutics
Locations (3):
- United States (3):
  - City of Hope, Duarte, California
  - Hackensack University Medical Center, Hackensack, New Jersey
  - MD Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: No